CLINICAL TRIAL: NCT05734664
Title: An Exploratory Clinical Study for the Development of a Novel Ultrasound Transducer Technology Intended for Non-invasive Monitoring of Cardiac Outputs
Brief Title: An Exploratory Clinical Study Non-invasive Monitoring of Cardiac Outputs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulsify Medical (Industry)
Collaborators: KU Leuven (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FIH_TechDemo1; CIV-22-03-03916 (Other: Eudamed)
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Output Measurements; Healthy Subjects
Keywords: Ultrasound Cardiac Non-invasive

STUDY DESIGN:
Intervention Model Description: Every subject will first undergo 2 scans with the Pulsify sensor. Immediately after acquisition with the Pulsify sensor, an echocardiographist will record a complete 2D and 3D ultrasound data set using a state-of-the-art equipment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scan with Pulsify sensor (Experimental): A trained operator will perform on each volunteer two scans with the Pulsify sensor. Both scans will have a different orientation of the sensor.
  Interventions: Device: Pulsify sensor
- Scan with state-of-the-art ultrasound equipment (Experimental): Immediately after acquisition with the Pulsify sensor, an echocardiographist will record a complete 2D and 3D ultrasound data set using a state-of-the-art equipment.
  Interventions: Device: State-of-the-art ultrasound equipment

INTERVENTIONS:
Device: Pulsify sensor — A positioning system will move the 1X1 cm Pulsify sensor step-by-step over a marked area of 10x10 cm on the subjects' chest to record a complete 3D data set of the heart. For accurate 3D reconstruction, the ECG and breathing cycle are also recorded during the acquisition using commercially available devices (Bitalino HeartBIT + Respiration Sensor). From the 3D dataset of the heart, the end-systolic and end-diastolic volumes will be extracted automatically to calculate the cardiac output.
  Arms: Scan with Pulsify sensor
Device: State-of-the-art ultrasound equipment — A complete 2D and 3D ultrasound data set using a GE Vivid E95 ultrasound machine, version 203 (General Electric Healthcare, Chicago, IL, United States) will be recorded. All data will be processed offline with a specialized software packet (EchoPAC, version 203, General Electric Healthcare, Chicago, IL, United States
  Arms: Scan with state-of-the-art ultrasound equipment

SUMMARY:
Pulsify Medical aims at developing a sensor designed for the non-invasive, continuous and real-time monitoring of cardiac hemodynamics in patients at risk based on new transducer technology and artificial intelligence. It relies on real-time 3D greyscale ultrasound reconstruction of the LV myocardium. This medical device is still under development and the main objective of this clinical investigation is to gather data on the accuracy of the current version of the sensor developed by Pulsify Medical to further guide the development of the device. The data generated will not be used for conformity assessment and this single-center prospective study on 8 patients is therefore deemed appropriate for this purpose.

During the pretreatment visit, eligibility of the subjects for the investigation will be assessed. Once subjects are considered eligible and they have consented to participate in the investigation, the visit to perform the monitoring will be scheduled. An operator will then perform on each patient two scans with the Pulsify sensor. For accurate 3D reconstruction, the ECG and breathing cycle during the acquisition will also be recorded. Immediately after acquisition with the Pulsify sensor, an echocardiographist will record a complete 2D and 3D ultrasound data set using regular ultrasound equipment used for medical examinations in the hospital. The data generated will then be used to compare the accuracy of the Pulsify sensor for cardiac output measurements with state-of-the-art ultrasound. The data will also enable to acquire a dataset of ultrasound images taken with the Pulsify sensor technology in a manner that is very close to the image capture mechanism of Pulsify's final product.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers can participate in this study if they:

* are aged over 18 years old
* have no known cardiovascular diseases
* are willing and able to comply with all investigation related procedures

Exclusion Criteria:

* Volunteers with arrhythmias, PM or ICD
* Volunteers with life supporting electronic devices (e.g. pacemakers)
* Volunteers with bad echocardiographic windows
* Volunteers post recent thorax surgery and open chest wounds
* Volunteers with abnormal thorax configuration (COPD, scoliosis, pectus excavatum, etc.) on criteria for the selection of topics
* Women in gestation
* Women that are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Comparison Cardiac Output | During procedure (1 hour)
  Compare the accuracy of the Pulsify sensor for cardiac output measurements with state-of-the-art ultrasound.

SECONDARY OUTCOMES:
Capture dataset | During procedure (1 hour)
  Acquire a dataset of ultrasound images taken with the Pulsify sensor technology in a manner that is very close to the image capture mechanism of Pulsify's final product. This dataset can be used for further image processing development.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Van De Bruaene, Principal Investigator — UZ Leuven; Lieven Herbots, Principal Investigator — Pulsify Medical
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
The investigational device is new and proprietary technology to Pulsify Medical. Data cannot be shared with others at the moment.